CLINICAL TRIAL: NCT03862963
Title: Lifestyle Intervention Trial to Treat Type 2 Diabetes in the Republic of the Marshall Islands
Brief Title: Lifestyle Intervention to Treat Diabetes in the Marshall Islands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Loma Linda University (Other); Brenda Davis Nutrition Consultation Services (Unknown); Canvasback Missions, Inc. (Unknown)
Responsible Party: Principal Investigator, Courtney M Peterson, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-170414009
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Parallel-arm study, although the control group was allowed to crossover after completing the control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Diabetes Care (Active Comparator): Standard of diabetes care in the Marshall Islands
  Interventions: Behavioral: Standard of diabetes care
- Lifestyle Intervention (Experimental): Plant-based, whole foods diet with moderate exercise
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Standard of diabetes care — The standard of diabetes care consisted of standard treatment protocols used by the MOH Diabetes Clinic. These included placing T2D patients on anti-hyperglycemic agents appropriate to their HbA1c levels (including sulfonylureas, metformin, and insulin) and providing oral and written information about the importance of maintaining a healthy weight, eating a healthy diet, and getting regular exercise. Participants in the control group were instructed not to make changes in their diet and activity levels during the study.
  Arms: Standard of Diabetes Care
Behavioral: Lifestyle Intervention — The lifestyle intervention consisted of a high-fiber, low-fat, mostly plant-based diet and 30-60 minutes per day of culturally-relevant, moderate intensity exercise. Participants initially received 12 weeks of group educational classes and some prepared meals and then followed the lifestyle intervention on their own for the remaining 12 weeks. Group classes included informative sessions on healthy eating, exercise (both aerobic and strength training), and stress management, as well as hands-on cooking classes. Classes were delivered as a combination of PowerPoint presentations, practical workshops, dine-outs, shopping tours, and cooking classes with spouses.
  Arms: Lifestyle Intervention

SUMMARY:
The Republic of the Marshall Islands has the highest prevalence of type 2 diabetes (T2D) in the world. This clinical trial tested whether a community-based, intensive, plant-rich lifestyle intervention with exercise is more effective for treating and managing T2D in the Republic of the Marshall Islands than the standard of diabetes care. The intensive lifestyle intervention consisted of a plant-rich diet and moderate exercise. It centered around a 12-week program of counseling and instruction on healthy eating, exercise, and stress management, as well as hands-on cooking classes and prepared meals. Cardiometabolic outcomes were assessed throughout the intervention and at 24 weeks. The present study is the first randomized clinical trial ever conducted in the Republic of the Marshall Islands and the first lifestyle intervention trial conducted in Micronesia.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the Republic of Marshall Islands
* Aged 18 - 75 years
* HbA1c ≥ 8.0% or diagnosed with T2D and taking diabetes medication
* Medical clearance to participate from Diabetes Wellness Center (DWC) physicians.

Exclusion Criteria:

* Recent (≤3 months) change in a diabetes-related medication dosage
* A physical or medical condition that would impede participation in the lifestyle intervention (e.g., wheel-chair bound, unstable angina)
* Evidence of significant coronary heart disease
* Previous participation in an intensive lifestyle intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2008-07-31

PRIMARY OUTCOMES:
Fasting glucose | Change from Week 0 to Week 24
  mg/dl
HbA1c | Change from Week 0 to Week 24
  Percent
Fasting insulin | Change from Week 0 to Week 24
  mU/l
HOMA-IR | Change from Week 0 to Week 24
  Insulin resistance as measured by HOMA-IR
Usage of diabetes medications | Change from Week 0 to Week 24
  Number as measured by the medication effect score

SECONDARY OUTCOMES:
Cholesterol (total, HDL, LDL) and triglycerides | Change from Week 0 to Week 24
  mg/dl
Blood pressure | Change from Week 0 to Week 24
  mm Hg
Heart rate | Change from Week 0 to Week 24
  beats/min
High-sensitivity C-reactive protein | Change from Week 0 to Week 24
  mg/l
Body weight | Change from Week 0 to Week 24
  kg
Body mass index (BMI) | Change from Week 0 to Week 24
  kg/m^2
Waist circumference | Change from Week 0 to Week 24
  cm

CONTACTS AND LOCATIONS:
Overall Officials: John H Kelly, M.D., Principal Investigator — Loma Linda University; Black Hills Lifestyle Medicine Center

REFERENCES:
- [Derived] Hanick CJ, Peterson CM, Davis BC, Sabate J, Kelly JH Jr. A whole-food, plant-based intensive lifestyle intervention improves glycaemic control and reduces medications in individuals with type 2 diabetes: a randomised controlled trial. Diabetologia. 2025 Feb;68(2):308-319. doi: 10.1007/s00125-024-06272-8. Epub 2024 Sep 21. PMID 39305340
- [Derived] Davis BC, Jamshed H, Peterson CM, Sabate J, Harris RD, Koratkar R, Spence JW, Kelly JH Jr. An Intensive Lifestyle Intervention to Treat Type 2 Diabetes in the Republic of the Marshall Islands: Protocol for a Randomized Controlled Trial. Front Nutr. 2019 Jun 5;6:79. doi: 10.3389/fnut.2019.00079. eCollection 2019. PMID 31231656